CLINICAL TRIAL: NCT06632834
Title: Outcome-targeted Therapy: Principle and Outcome Evaluation: Clinical Study, and Phenotype-genotype Correlation
Brief Title: Outcome-targeted Therapy: Principle and Outcome Evaluation: Clinical Study and Phenotype-genotype Correlation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201912067MINB
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dilated Cardiomyopathy
Keywords: cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: 1. A retrospective and prospective cohort study will be conducted. Patients diagnosed with DCM below the age of 35 years from 1990 to 2019 will be enrolled. Medical records will be reviewed. A 3-stage genetic testing will be performed after informed consent.
  2. An open-labeled, exploratory study of simvastatin on the cardiac function of DCM patients will be conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simvastatin (Experimental): Simvastatin added with baseline anti-congestive medication in dilated cardiomyopathy patient.
  Interventions: Drug: simvastatin therapy

INTERVENTIONS:
Drug: simvastatin therapy — Simvastatin should be administered initially with the dose of 10 mg once daily for adult and 0.25 mg/Kg once daily for children. Dose of simvastatin will be increased to the dose of 20 mg once daily for adult and 0.5 mg/Kg once daily for children after the check at 3 months without adverse effects.

SUMMARY:
Brief Summary(Use lay language. Include a statement of the study hypothesis.):

Dilated cardiomyopathy (DCM) is the most common childhood cardiomyopathy and is associated with significant early morbidity and mortality. Those who fail to improve within the first year of diagnosis usually deteriorated even upon aggressive anti-congestive medications. Investigators had conducted precision-medicine-based approach to provide strategic approach as drug repurposing to identify new treatments. Investigators have identified the beneficial effects from a statin, simvastatin, to restore the cardiac contractility in the human induced pluripotent stem cell lines derived from a DCM proband and the proband's father. The mutant mouse consequently confirmed the beneficial effects. The initial experience in the proband is promising. This clinical trial is to find out if simvastatin will benefit the cardiac function of DCM patients.

DETAILED DESCRIPTION:
Dilated cardiomyopathy (DCM) is the most common childhood cardiomyopathy and is associated with significant early morbidity and mortality. About half of patients die or require heart transplantation within 5 years of diagnosis. The survival advantage from transplantation is limited, particularly in DCM infants.The medical therapy for DCM with heart failure includes anti-congestive medications and antiplatelet therapy. Those who fail to improve within the first year of diagnosis usually deteriorated even upon aggressive anti-congestive medications. Investigators have conducted precision-medicine-based approach to provide strategic approach as drug repurposing to identify new treatments. Investigators have identified the beneficial effects from a statin, simvastatin, to restore the cardiac contractility in the human induced pluripotent stem cell lines derived from a DCM proband and the proband's father. The mutant mouse consequently confirmed the beneficial effects. The initial experience in the proband is promising. The proband was diagnosed as DCM with severe heart failure during infancy. Family screening identified that the proband's father had dilated left ventricle (LV) and low LV ejection fraction (LVEF). Genetic examination of this DCM family revealed that the proband and the proband's father had heterogeneous missense mutation. About 2 years after the disease onset, participants growth was slow, the LVEF remained poor and the NT-pro BNP level was high under aggressive anti-congestive medications. Because of the beneficial effects of simvastatin from in vitro study and in vivo animal study, off-label use of simvastatin was initiated after obtaining the parents' agreement. Participants general condition and cardiac condition 4 years after the disease onset and 1.5 years after the simvastatin therapy improved without adverse effects. The LVEF increased from 17.5% to 39.2% and the NT-pro BNP level dropped from 1200 to 363 pg/ml. Simvastatin is effective in lowing LDL and cholesterol, thereby to improve the outcome of patients with coronary arterial disease, familiar hypercholesterolemia, etc. For children, though the dosage range and the indication remain unclear, it had been used in children with various diseases. Simvastatin had been given in a small cohort of adult DCM. Patients treated with simvastatin had a lower New York Heart Association functional class compared with those receiving placebo. The LVEF also improved in the simvastatin group. This clinical trial is to find out if simvastatin will benefit the cardiac function of DCM patients.

ELIGIBILITY:
Inclusion criteria

Patients diagnosed as dilated cardiomyopathy, classified as NYHA functional class II or III and still have a low left ventricular ejection fraction (LVEF) (LVEF < 45% and the Z score of the LV end-diastolic diameter > 2.0) will be enrolled, if they have normal or high level of cholesterol and triglyceride and fulfill any of the following criteria:

1. Patients who have already received anti-congestive medications for at least three months and still have poor LV function (LVEF < 45% and the Z score of the LV end-diastolic diameter > 2.0).
2. Patients who have persistent or even worsening heart failure after one month of anti-congestive medications.
3. Patients who have positive family history of dilated cardiomyopathy and have received anti-congestive medications for one month.
4. Patients or their parents must sign an informed consent form.

Exclusion criteria

Patients who fulfill any of the following criteria will be excluded from the trial:

1. Patients who underwent prior cardiac surgery. Those who received DCM related surgery, such as mitral valve plasy, for longer than a year are not subject to this restriction.
2. Patients who had active liver / renal dysfunction.
3. Concomitant use with gemfibrozil, cyclosporine, danazol, strong CYP3A4 inhibitors (eg, boceprevir, clarithromycin, erythromycin, HIV protease inhibitors, itraconazole, ketoconazole, nefazodone, posaconazole, telaprevir, telithromycin, voriconazole), or cobicistat-containing products
4. Patients who are pregnant or plan to pregnancy in the period of study.
5. Patients who are intolerance to simvastatin therapy.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2025-01-19 (Estimated); Study Completion 2025-01-19 (Estimated)

PRIMARY OUTCOMES:
Improvement in left ventricular ejection fraction and NT-pro BNP (biomarker for left ventricular function)) | 2 years
  The changes from baseline to completion of the study in the echocardiographic parameters for LV function, the left ventricular ejection fraction.The changes in the biomarker for left ventricular function(pro-BNP) from baseline to completion of the study will be evaluated by a repeated assessment.
  Preliminary data
  Our preliminary data from pediatric DCM population showed that the 1-year-, and 5-year transplant-free survival after diagnosis were 61.3%, and 45.2%. None of infant patients received heart transplant and the waitlist mortality were high.
  The proband patient was diagnosed as DCM at the age of 6 months. Two years after the diagnosis, participants cardiac condition was stagnant. Because of the beneficial effects of simvastatin from in vitro and in vivo animal study, off-label use was initiated after obtaining the parents' agreement. Participants LVEF increased from 17.5% to 42% and the NT-pro BNP level dropped from 1200 to 217 pg/ml.

SECONDARY OUTCOMES:
Progression free survival and overall survival | 2 years
  Progression-free survival is measured from the date of starting treatment to the date of disease progression (increase of LVEF for 6% or prior pro-BNP for 10%), to death without progression, or to the last follow-up without progression.Overall survival is measured from the date of starting treatment in the study to the date of death, or to the last follow-up without death.Safety variables include toxicity grading, adverse events, and laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chieh Tseng, MD, Principal Investigator — Principal Investigator
Locations (1):
- National Taiwan University Hospital, Taipei County, Zhongzheng District, Taiwan